CLINICAL TRIAL: NCT06988280
Title: Ultrasound-guided Transvaginal Aspiration of Cystic Pelvic Lesions
Acronym: UTAC
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S68671
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-03

CONDITIONS: Pelvic Abscess; Adnexal Cyst; Ovarian Neoplasms
Keywords: adnexal cyst; transvaginal aspiration; cyst recurrence; pelvic abscess; symptom relief
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pelvic cystic lesions (i.e adnexal lesions and abscesses): Patients with cystic lesions (i.e adnexal lesions and abscesses), undergoing an ultrasound-guided transvaginal drainage as per our standard of practice.
  Interventions: Diagnostic Test: Ultrasound-guided transvaginal aspiration of cystic pelvic lesions.

INTERVENTIONS:
Diagnostic Test: Ultrasound-guided transvaginal aspiration of cystic pelvic lesions. — Ultrasound-guided transvaginal aspiration is a minimally invasive procedure used to drain cystic pelvic lesions, such as adnexal cysts or pelvic abscesses. A thin needle is inserted through the vaginal wall under ultrasound guidance to aspirate fluid from the cyst, reducing its size.

SUMMARY:
Adnexal cysts or pseudocysts are a common finding on transvaginal ultrasound, especially in premenopausal women. Due to the size of some cysts, they may cause discomfort. Moreover, a genuine risk of ovarian torsion presents when these lesions grow.

During the last decades, great advancements have been made in the correct differentiation of benign from malignant lesions. However, there still is controversy concerning the optimal treatment approach of symptomatic adnexal cysts with a low risk of malignancy, consisting of both surgery or ultrasound-guided transvaginal aspiration. Factors such as comorbidities and lesion characteristics need to be considered when counselling patients, as well as the possibility of short term recurrence.

Surgically removing them may result in longer hospital stays and recovery, with higher costs, while transvaginal needle aspiration techniques can be performed during a consultation. Additional benefits in avoiding surgery, particularly in women of reproductive age, are fertility preservation and less pelvic adhesions.

On the other hand, the main arguments against cyst aspiration are the relatively high recurrence rate of cysts, the minimal risk of malignant cell dissemination (In case of a false negative diagnosis) and the cytological instead of a histopathological examination.

With this in mind, it is important to base management decisions on the sonographic features of the lesions.

In addition, cyst aspiration can also be considered in large symptomatic cysts with a high risk of malignancy, but where curative treatment with surgical or chemotherapeutical intervention cannot be considered due to poor general condition of the patient. Especially in the absence of large volume ascites or peritoneal carcinomatosis, but with significant symptoms due to lesion size, cyst aspiration may give short term symptom alleviation. Given the risk of cancer cell dissemination, this intervention is always discussed in a multidisciplinary team discussion, to balance risk and benefits for patients with no other treatment options, Transvaginal needle aspiration is also being used in pelvic abscesses. The study of K. Gjelland et al. found that transvaginal aspiration combined with antibiotic treatment of pelvic abscesses is equally effective as surgically removing them. They state that this should be first-line treatment for abscesses, as it is minimally invasive, leading to better patient tolerance and avoiding the risks associated with anesthesia and surgery.

Saline irrigation of the abscess cavity can be performed, making the process of pus aspiration easier when the consistency is too viscous.

The literature still lacks studies about the symptom relief in patients receiving treatment for pelvic cystic lesions. Given that this is an important outcome parameter in determining the feasibility of performing procedures, more research in this area is needed.

The main aim of this prospective study is to evaluate the patient's symptom relief and cyst recurrence rate after ultrasound-guided transvaginal aspiration of pelvic cystic lesions or abscess drainage. Secondly, the safety and the patient's overall experience during as well as immediately after the procedure will be assessed.

ELIGIBILITY:
Participants eligible for inclusion in this study must meet all of the following criteria:

1. Lesion criteria applicable for therapeutic intervention

   1. Safe accessibility of the lesion (within reach of aspiration needle; visible on ultrasound; transvaginal access; no interposition of bowel or blood vessels)
   2. Lesion types included: cystic lesions (adnexal cysts), pelvic inclusion cysts (pseudocysts), pelvic abscesses
2. Indications

   1. Pain relief in symptomatic cystic lesions with benign appearance.
   2. Symptomatic treatment in probably malignant lesions (only in non-curative setting).

Exclusion Criteria:

1. Patients <18 years
2. Poor performance status contra-indicating the procedure
3. Vaginal stenosis (severe atrophy - virgo - vaginismus)
4. Purely solid lesions
5. Cystic lesions with a presumed malignant diagnosis and a risk of tumor dissemination in a curative setting
6. Physiological cysts in asymptomatic patients (in case of doubt the patient is reassessed after 3-6 months)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients elligible based on the above mentioned criteria in University Hospitals Leuven.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pain on verbal rating scale (0-10) | • Pain scores indicated by the patient prior to the procedure, during the procedure, one week after and three months after the procedure (based on a verbal rating scale).
  Pain scores indicated by the patient prior to the procedure, during the procedure, one week after and three months after the procedure.
Recurrence of cyst (binary outcome after 12 months) | 12 months
  Clinical and sonographic follow-up of possible recurrence (up till 12 months). Routine assessment will be done after 3 and 12 months

SECONDARY OUTCOMES:
General experience during the procedure (based on verbal rating scale 0-10) | Right after the procedure to 3 days after.
  General experience during the procedure based on verbal rating scale, assessed after the procedure by an independent examiner.
Complications (based on Clavien Dindo classification) | Immediately after the procedure to 6 weeks after the procedure.
  Registration of adverse events, such as Vasovagal reaction, bleeding, infection, excessive pain.

OTHER OUTCOMES:
Cytological and possible microbial analysis of the aspirate. | From the procedure (enrollment) to 2 weeks after the procedure.
  Assessment of cytological and microbiological analysis of the aspirate if relevant.
Difference of inflammatory markers (White blood cell count) | From the procedure (enrollment) to 2 weeks after the procedure.
  Only applicable in presumed pelvic abscess; Measured at the time of the procedure and 48 hours later, as per our standard ofpractice.
Difference in inflammatory markers (C-reactive protein) | From the procedure (enrollment) to 2 weeks after the procedure.
  Only applicable in presumed pelvic abscess; Measured at the time of the procedure and 48 hours later, as per our standard ofpractice.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be added in the journal submission, and will be made available to other investigators on reasonable request.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Saokar A, Arellano RS, Gervais DA, Mueller PR, Hahn PF, Lee SI. Transvaginal drainage of pelvic fluid collections: results, expectations, and experience. AJR Am J Roentgenol. 2008 Nov;191(5):1352-8. doi: 10.2214/AJR.07.3808. PMID 18941068
- [Background] Feld R, Eschelman DJ, Sagerman JE, Segal S, Hovsepian DM, Sullivan KL. Treatment of pelvic abscesses and other fluid collections: efficacy of transvaginal sonographically guided aspiration and drainage. AJR Am J Roentgenol. 1994 Nov;163(5):1141-5. doi: 10.2214/ajr.163.5.7976890.
- [Background] Caspi B, Goldchmit R, Zalel Y, Appelman Z, Insler V. Sonographically guided aspiration of ovarian cyst with simple appearance. J Ultrasound Med. 1996 Apr;15(4):297-300. doi: 10.7863/jum.1996.15.4.297. PMID 8683664
- [Background] Troiano RN, Taylor KJ. Sonographically guided therapeutic aspiration of benign-appearing ovarian cysts and endometriomas. AJR Am J Roentgenol. 1998 Dec;171(6):1601-5. doi: 10.2214/ajr.171.6.9843295.
- [Background] Corsi PJ, Johnson SC, Gonik B, Hendrix SL, McNeeley SG Jr, Diamond MP. Transvaginal ultrasound-guided aspiration of pelvic abscesses. Infect Dis Obstet Gynecol. 1999;7(5):216-21. doi: 10.1002/(SICI)1098-0997(1999)7:53.0.CO;2-N. PMID 10524665
- [Background] Gjelland K, Ekerhovd E, Granberg S. Transvaginal ultrasound-guided aspiration for treatment of tubo-ovarian abscess: a study of 302 cases. Am J Obstet Gynecol. 2005 Oct;193(4):1323-30. doi: 10.1016/j.ajog.2005.06.019. PMID 16202721
- [Background] Urfali FE, Korkmaz M, Zeren S, Yaylak F, Tok Umay S. Percutaneous drainage as an rapid procedure for deep pelvic abscess in the emergency department. Ulus Travma Acil Cerrahi Derg. 2021 Sep;27(5):534-538. doi: 10.14744/tjtes.2020.99478. PMID 34476798
- [Background] Tsai CC, Shen CC, Changchien CC, Hsu TY, Kung FT, Chang SY, Chang MY, Huang FJ. Ultrasound-guided transvaginal cyst aspiration for the management of pelvic pseudocyst: a preliminary experience. Chang Gung Med J. 2002 Nov;25(11):751-7. PMID 12553363
- [Background] Timmerman D, Van Calster B, Testa A, Savelli L, Fischerova D, Froyman W, Wynants L, Van Holsbeke C, Epstein E, Franchi D, Kaijser J, Czekierdowski A, Guerriero S, Fruscio R, Leone FPG, Rossi A, Landolfo C, Vergote I, Bourne T, Valentin L. Predicting the risk of malignancy in adnexal masses based on the Simple Rules from the International Ovarian Tumor Analysis group. Am J Obstet Gynecol. 2016 Apr;214(4):424-437. doi: 10.1016/j.ajog.2016.01.007. Epub 2016 Jan 19. PMID 26800772
- [Background] Duke D, Colville J, Keeling A, Broe D, Fotheringham T, Lee MJ. Transvaginal aspiration of ovarian cysts: long-term follow-up. Cardiovasc Intervent Radiol. 2006 May-Jun;29(3):401-5. doi: 10.1007/s00270-005-0167-0. PMID 16502175
- [Background] Diaz de la Noval B, Rodriguez Suarez MJ, Fernandez Ferrera CB, Valdes Lafuente D, Arias Cailleau R, Perez Arias H, Torrejon Becerra JC, Suarez Gil P, Lucio Gonzalez LR. Transvaginal Ultrasound-Guided Fine-Needle Aspiration of Adnexal Cysts With a Low Risk of Malignancy: Our Experience and Recommendations. J Ultrasound Med. 2020 Sep;39(9):1787-1797. doi: 10.1002/jum.15283. Epub 2020 Apr 16. PMID 32298023
- [Background] Garcia-Tejedor A, Castellarnau M, Burdio F, Fernandez E, Marti D, Pla MJ, Ponce J. Ultrasound-guided aspiration of adnexal cysts with a low risk of malignancy: is it a recommendable option? J Ultrasound Med. 2015 Jun;34(6):985-91. doi: 10.7863/ultra.34.6.985. PMID 26014317
- [Background] Kostrzewa M, Zajac A, Wilczynski JR, Stachowiak G. Retrospective analysis of transvaginal ultrasound-guided aspiration of simple ovarian cysts. Adv Clin Exp Med. 2019 Nov;28(11):1531-1535. doi: 10.17219/acem/104549. PMID 31660708